CLINICAL TRIAL: NCT07306364
Title: Psilocybin in Chronic Low Back Pain: An Integrative Study of Lab-Based Mechanisms and Real-World Physical Therapy Outcomes
Brief Title: Psilocybin-Assisted Physical Therapy in Chronic Low Back Pain
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Joao De Aquino, Assistant Professor of Psychiatry, Yale University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2000041668
Record Dates: First submitted 2025-12-23; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Chronic Low Back Pain (CLBP); Physical Therapy; Psilocybin
MeSH Terms: interventions — Psilocybin; Niacin

STUDY DESIGN:
Intervention Model Description: Adults with CLBP beginning a course of PT will be allocated equally into three parallel arms. Participants will receive a single oral dose of either low-dose psilocybin (10 mg), moderate-dose psilocybin (25 mg), or placebo (niacin). All three groups will follow identical study procedures.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Low-dose psilocybin (10 mg) (Active Comparator)
  Interventions: Drug: Psilocybin 10 mg
- Moderate-dose psilocybin (25 mg) (Active Comparator)
  Interventions: Drug: Psilocybin 25 mg
- Placebo (niacin). (Placebo Comparator)
  Interventions: Drug: Niacin 100 mg

INTERVENTIONS:
Drug: Psilocybin 10 mg — Two 5 mg psilocybin capsuels will be administered to participants randomized into the low-dose psilocybin group.
  Arms: Low-dose psilocybin (10 mg)
Drug: Psilocybin 25 mg — One 25 mg psilocybin capsuel and one 100 mg niacin (placebo) capsuel will be administered to participants radomized into the moderate-dose psilocybin group.
  Arms: Moderate-dose psilocybin (25 mg)
Drug: Niacin 100 mg — Two 100 mg niacin capsuels will be adminstered to participants randomized to the placebo group.
  Arms: Placebo (niacin).

SUMMARY:
The purpose of this research study is to investigate whether a single administration of psilocybin can improve interoceptive awareness (awareness of bodily sensations) in individuals with chronic low back pain undergoing physical therapy, and whether these improvements are linked to pain relief and better physical therapy outcomes.

DETAILED DESCRIPTION:
Preclinical and human studies suggest that psilocybin can temporarily disrupt rigid, maladaptive patterns of brain activity and promote longer-lasting changes in how the brain processes internal sensations. People with chronic pain who have used psilocybin qualitatively describe feeling more aware of their bodies, able to reinterpret pain sensations, and less distressed and disabled by their pain.

Building on these mechanistic insights, this randomized, double-blind, placebo-controlled trial will evaluate a single dose of low- (10 mg), moderate-dose (25 mg), or placebo (niacin) administered prior to a standardized course of physical therapy (PT) in adults with chronic low back pain (CLBP). Participants in both treatment groups will receive a course of PT that is consistent with what would be delivered outside of involvement in the research study. That is, the study is evaluating psilocybin as an adjunct to PT delivered in a community outpatient PT clinic. By testing whether psilocybin-induced recalibration of brain networks can enhance engagement with and outcomes of PT, this study aims to establish a novel, non-opioid integrative strategy to relieve CLBP and restore functional recovery.

ELIGIBILITY:
Inclusion Criteria:

* 1. Ability to provide informed consent in English.
* 2. Provision of signed and dated informed consent form.
* 3. Stated willingness to comply with all study procedures and availability for the duration of the study.
* 4. Male and female participants aged 18-65 years.
* 5. CLBP, uniformly defined as high-impact or bothersome non-cancer low back pain lasting ≥ three months that occurs most days and limits life or work activities.
* 6. At least moderate pain-related disability as measured by a total score on the ODI ≥ 15.
* 7. For women of childbearing potential, must have a negative urine pregnancy test at screening and immediately before dose administration.

  * Negative urine pregnancy test at screening and immediately before dose administration.
  * Use of one highly effective contraception (e.g., IUD, barrier method) for ≥ 1 month prior to screening.
* 8. Participants are required to commit to employing dual contraceptive methods throughout the study and to abstain from sperm or egg donation during the study period and for 28 days following the final drug dose for ova, and for 90 days following the final drug dose for sperm. Dual contraceptive methods encompass the use of a barrier contraceptive, such as condoms, coupled with another effective method capable of preventing pregnancy, such as oral or parenteral contraceptives, intrauterine devices, spermicide, and the like.
* 9. Resting blood pressure ≤ 140/90 mmHg (average of three screenings) and resting heart rate 60-100 bpm.
* 10. Normal screening EKG: QTcF < 450 ms; no clinically significant arrhythmias, ischemia, or bundle branch block.
* 11. Hepatic and renal function within acceptable limits: AST/ALT ≤ 2× ULN; bilirubin ≤ 1.5× ULN; eGFR ≥ 50 mL/min/1.73 m².
* 12. Ability to safely ingest oral capsules for the dosing visit.
* 13. Safe transportation plan after the dosing session (e.g., designated driver).
* 14. Signed medical release permitting the study team to communicate with outside providers for medication/therapy history or crisis management.
* 15. Designation of an adult emergency contact (relative, spouse, close friend) willing to monitor for mood/behavior changes post-dose and provide transportation if needed.
* 16. Agreement to attend preparatory and integration sessions, follow-up visits, and to respond to telephone/email contacts.

Exclusion Criteria:

* 1. Hallucinogen Use Disorder or Hallucinogen Persisting Perceptual Disorder.
* 2. Personal or family history of schizophrenia, schizoaffective disorder, bipolar disorder, or major depressive disorder with psychotic features; any history of substance-induced psychosis or current psychotic symptoms at Screening per the Brief Psychiatric Rating Scale.
* 3. Active suicidal ideation or behavior in the past 3 months, as indicated on the C-SSRS.
* 4. Lifetime use of classic psychedelics (5-HT2A agonists) within the preceding 12 months, or unwillingness to abstain from their use for up to 4 weeks post-dose.
* 5. Current moderate or severe depression, as indicated by a score of ≥ 3 on the depression subscale (items 1 and 2) of the Patient Health Questionnaire-4 (PHQ-4).
* 6. Total score on the ODI ≥ 35, indicating an individual is "completely disabled."
* 7. Meeting DSM-5 criteria for alcohol or substance use disorders (other than tobacco use disorder) within the last year; use of THC-containing products > 2×/week over the past 30 days or unwillingness to abstain for at least 1 week pre-dose through 4 weeks post-dose. Abstinence will be confirmed via point-of-care urine 11-nor-9-carboxy-THC testing with a cut-off ≤ 50 ng/mL.
* 8. Clinically significant medical disorders (e.g., moderate-to-severe hepatic impairment [Child-Pugh B/C], AST/ALT > 2× ULN, bilirubin > 1.5× ULN, eGFR < 50 mL/min/1.73 m², diabetes, uncontrolled thyroid disease).
* 9. Neurological conditions altering nociceptive response (e.g., stroke, neuropathy) or history of seizure/head injury with > 30 minutes loss of consciousness.
* 10. Contraindications to nociceptive testing (e.g., untreated hypertension > 140/90 mmHg).
* 11. Current use of serotonergic medications (e.g., SSRIs, SNRIs, TCAs).
* 12. Current regular use of medications affecting pain (e.g., opioids, gabapentinoids, cyclobenzaprine).
* 13. Current regular use of inhibitors of UGT1A9, UGT1A10, MAO and aldehyde or alcohol dehydrogenase.
* 14. Major neurocognitive disorders (e.g., dementia) or any cognitive deficit impairing consent/participation.
* 15. Abnormal EKG findings (e.g., ischemia, infarct patterns, bundle branch block, atrial fibrillation, QTcF ≥ 450 ms).
* 16. Resting QTcF prolongation or other torsades de pointes risk factors (uncontrolled electrolyte disturbances, family history of sudden death, torsadogenic medications).
* 17. Any other condition that, in the investigator's judgment, would compromise safety or ability to complete the study.
* 18. Known or suspected cardiovascular disease, including but not limited to atrial fibrillation, coronary artery disease, history of myocardial infarction, structural heart disease, congestive heart failure, or uncontrolled hypertension.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2029-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Change in interoceptive awareness as measured by the Multidimensional Assessment of Interoceptive Awareness-2 from 4 weeks post-dose to 8 weeks post dose | 4 weeks post dose, 8 weeks post-dose
  The Multidimensional Assessment of Interoceptive Awareness-2 (MAIA-2) is a validated 37-item, self-report instrument assessing mind-body connections (i.e., interoceptive awareness). MAIA-2 scoring involves rating the 37 items on a 0 (never) to 5 (always) Likert scale, resulting in scores for eight subscales (Noticing, Not-distracting, Not-worrying, Attention regulation, Emotional awareness, Self-regulation, Body Listening, Trusting). Scores for each of the 8 scales are averaged (sum of items divided by number of subscale items). Higher scores indicate better interoceptive awareness. Change = (8-week post-dose score - 4-week post-dose score).
Change in Pain, Enjoyment, and General Activity (PEG) total score at 8 weeks post dose | 4 weeks post-dose, 8 weeks post-dose
  The Pain, Enjoyment, General Activity (PEG) Scale is a 3-item questionnaire used to measure how chronic pain affects a person's life, focusing on average pain intensity (P), interference with enjoyment (E), and interference with general activity (G) using 0-10 Likert scale for each item. The final PEG score is calculated by adding the three scores and dividing by three. Scores range from 0-10, with higer scores indicating higher pain impact. Change= (8-week post-dose score - 4-week post-dose score).
Change in functional disability measured by the Oswestry Disability Index (ODI) from baseline to 8 weeks post-dose. | Baseline (Day 0), 8 weeks post-dose
  The Oswestry Disability Index (ODI) is a widely used, 10-question self-report questionnaire that measures functional disability and quality of life for people with low back pain, assessing activities like walking, sitting, sleeping, and pain intensity, with scores ranging from 0-100% categorized into minimal (0-20%), moderate (21-40%), severe (41-60%), crippled (61-80%), and bed-bound (81-100%) disability. Change = (8-week post-dose score - baseline [day 0] score)

SECONDARY OUTCOMES:
Physical activity measured by average daily step count via daily Experience Sampling Monitoring (ESM) | Daily for approximately 28 days post-dose
  Participants will record their daily step count via study-provided pedometer from 4 weeks post dose to 8 weeks post-dose. The average step count will be assessed.
Change in functional mobility from 4 weeks post-dose to 8 weeks post-dose measured by the 10-Meter Walk Test (10MWT) | 4 weeks post-dose, 8 weeks post-dose
  The 10-Meter Walk Test (10MWT) is a common physical therapy assessment measuring how fast someone walks over a short distance, typically 10 meters. The 10MWT will be used to evaluate gait velocity. Change= (8-week post dose score - 4-week post-dose score)
Change in functional mobility from 4 weeks post-dose to 8 weeks post-dose measured by the 30-Second Sit to Stand (30STS) | 4 weeks post-dose, 8 weeks post-dose
  The 30 Second Sit to Stand Test (30STS) is a common physical therapy assessment recording the number of times a person can stand from a chair over 30 seconds. The 30STS will evaluate functional lower extremity strength and endurance. Change= (8-week post dose score - 4-week post-dose score).
Change in back-specific strength from 4 weeks post-dose to 8 weeks post-dose, measured by myotomal dynamometry spanning vertebrae L2 to S2 using an isometric deadlift test. | 4 weeks post-dose, 8 weeks post-dose
  Myotomal dynamometry spanning vertebral levels L2-S2 will be performed by testing the muscle groups associated with each spinal nerve root using a handheld dynamometer or graded manual resistance. Change scores will be calculated as: 8-week post-dose value minus 4-week post-dose value
Nociceptive sensitivity assessed by a composite multimodal Quantitative Sensory Testing (QST) battery | 4 weeks post-dose, 8 weeks post-dose
  Quantitative sensory testing (QST) will assess multiple pain modalities including pressure, thermal, and cold pressor, pain threshold and tolerance; Mechanical temporal summation; Thermal temporal summation; and Conditioned pain modulation. All raw QST values will be converted to standardized Z-scores. A general pain sensitivity score will be derived by averaging the Z-scores for pressure pain threshold, heat pain threshold, heat pain tolerance, and cold pressor latency; higher scores indicate greater overall pain sensitivity. Central sensitization will be quantified by averaging the Z-scores for mechanical temporal summation, thermal temporal summation, conditioned pain modulation, and after-sensation ratings; positive values reflect a pronociceptive state, while negative values indicate an antinociceptive state.
Fear of movement measured using the physical activity subscale of the Fear Avoidance Beliefs Questionnaire (FABQ-PA) mean score | 4 weeks post-dose, 8 weeks post-dose
  The Fear Avoidance Beliefs Questionnaire (FABQ-PA) is a 5-item subscale of the broader FABQ, used to measure how much a person's fear of pain makes them believe physical activity will worsen their condition, leading to avoidance. Responses are rated from 0 (completely disagree) to 6 (completely agree) for a maximum of 24 points. A score of 15 or higher often signifies significant fear-avoidance beliefs about physical activity.
Pain catastrophizing measured by the Pain Catastrophizing Scale (PCS-6) and Situational Catastrophizing Questionnaire (SCQ) mean score | 4 weeks post-dose, 8 weeks post-dose
  The Pain Catastrophizing Scale (PCS-6) is a 6-item version of the Pain Catastrophizing Scale (PCS), designed to quickly measure negative thinking about pain (rumination, magnification, helplessness). The PCS-6 is scored on a Likert scale with values from 0 ("Not at all") to 4 ("All the time"). Scores range from 0-24, with higher scores indicating greater pain catastrophizing.
Situational pain catastrophizing measured by the Situational Catastrophizing Questionnaire (SCQ) mean score | 4 weeks post-dose, 8 weeks post-dose
  The Situational Catastrophizing Questionnaire consists of 6 items that assess negative thoughts and feelings in response to a specific pain stimulus. The SCQ is scored on a Likert scale with values from 0 ("Not at all") to 4 ("All the time"). Scores range from 0-24, with higher scores indicating greater negative thoughts and feelings. The SCQ will be asseesed after participants complete the QST battery.
Daily pain intensity/interference measured by the Pain, Enjoyment, General Activity (PEG) Scale via daily Experience Sampling Monitoring (ESM) mean score | Daily for approximitely 28 days post-dose
  The Pain, Enjoyment, General Activity (PEG) Scale is a 3-item questionnaire used to measure how chronic pain affects a person's life, focusing on average pain intensity (P), interference with enjoyment (E), and interference with general activity (G) using 0-10 Likert scale for each item. The final PEG score is calculated by adding the three scores and dividing by three. Scores range from 0-10, with higer scores indicating higher pain impact. Participants will complete the PEG Scale daily via ESM from 4 weeks post dose to 8 weeks post-dose.
Daily pain affect measured by the Positive and Negative Affect Schedule (PANAS) via daily Experience Sampling Monitoring (ESM) mean score | Daily for approximitely 28 days post-dose
  the Positive and Negative Affect Schedule (PANAS) is a 20-item self-report questionnaire listing adjectives relating to Positive Affect (PA) (e.g., excited, inspired) and Negative Affect (NA) (e.g., distressed, afraid). Items are rated on a Likert scale ranging from 1 "Very slightly or not at all" to 5 "extremely". The PANAS yeilds separate PA and NA scores, each ranging from 10 to 50. Higher PA scores indicate more positive feelings, while higher NA scores indicate more negative feelings. These scores are used to track emotional states over time.
  Participants will complete the PANAS daily via ESM from 4 weeks post dose to 8 weeks post-dose.
Psychedelic-related adverse events will be measured by the Swiss Psychedelic Side Effect Inventory (SPSI) | 8 hours post-dose
  The Swiss Psychedelic Side Effect Inventory (SPSI) is a standardized 32-item questionnaire designed for the systematic assessment and recording of adverse effects from psychedelics. For each reported side effect, the SPSI assesses: Severity (light, moderate, strong), Duration, Impact (from very disadvantageous to very advantageous), and Treatment-relatedness. Number of The number of participants, in each group, experiencing at least one event on the SPSI will be tabulated by event frequency and severity and summarized in descriptive tables.
Subjective psychedelic effects will be measured by the 5-Dimensional Altered States of Consciousness Scale (5D-ASC) mean score | 8 hours post-dose
  The 5-Dimensional Altered States of Consciousness Scale (5D-ASC) is a 94-item self-report questionnaire used to quantify participants subjective experiences of altered states of consciousness induced by psychedelics. Items are rated using a 100-millimeter visual analogue scale (VAS), indicating to what extent the experience applied to them during or after a specific event (e.g., from "No, not more than usually" to "Yes, very much more than usually"). The 5D-ASC is divided into 11 subscales: Oceanic Boundlessness, Anxious Ego Dissolution, Visionary Restructuralization, Auditory Alterations, Reduction of Vigilance. The scores within each subscale are averaged to produce a mean score for that specific subscale or dimension. Descriptives for the 5D-ASC will be tabulated by event frequency and severity and summarized in descriptive tables.

OTHER OUTCOMES:
Peak Plasma Concentration (Cmax) of Psilocybin | 30 minutes pre-dose; 60, 120, 240, and 360 minutes post-dose
  Plasma psilocybin concentrations (Units: ng/mL) will be measured at pre-dose (-30 minutes) and at 60, 120, 240, and 360 minutes post-dose. Cmax (peak observed plasma concentration) of psilocybin will be derived from these timepoints using noncompartmental methods.
Area Under the Plasma Concentration-Time Curve from 0 to 6 Hours (AUC0-6h) of Psilocybin | 30 minutes pre-dose; 60, 120, 240, and 360 minutes post-dose
  Plasma psilocybin concentrations will be measured at pre-dose (-30 minutes) and at 60, 120, 240, and 360 minutes post-dose. AUC0-6h for psilocybin will be calculated using noncompartmental analysis (e.g., trapezoidal rule) over the 0-6 hour post-dose period.
Peak Plasma Concentration (Cmax) of Psilocin | 30 minutes pre-dose; 60, 120, 240, and 360 minutes post-dose
  Plasma psilocin concentrations (ng/mL) will be measured at pre-dose (-30 minutes) and at 60, 120, 240, and 360 minutes post-dose. Cmax (peak observed plasma concentration) of psilocin will be derived from these timepoints using noncompartmental methods.
Area Under the Plasma Concentration-Time Curve from 0 to 6 Hours (AUC0-6h) of Psilocin | 30 minutes pre-dose; 60, 120, 240, and 360 minutes post-dose
  Plasma psilocin concentrations will be measured at pre-dose (-30 minutes) and at 60, 120, 240, and 360 minutes post-dose. AUC0-6h for psilocin will be calculated using noncompartmental analysis (e.g., trapezoidal rule) over the 0-6 hour post-dose period.

CONTACTS AND LOCATIONS:
Overall Officials: Joao De Aquino, M.D., Principal Investigator — Yale University
Locations (1):
- Connecticut Mental Health Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bornemann J, Close JB, Spriggs MJ, Carhart-Harris R, Roseman L. Self-Medication for Chronic Pain Using Classic Psychedelics: A Qualitative Investigation to Inform Future Research. Front Psychiatry. 2021 Nov 12;12:735427. doi: 10.3389/fpsyt.2021.735427. eCollection 2021. PMID 34867525
- [Background] Skosnik PD, Sloshower J, Safi-Aghdam H, Pathania S, Syed S, Pittman B, D'Souza DC. Sub-acute effects of psilocybin on EEG correlates of neural plasticity in major depression: Relationship to symptoms. J Psychopharmacol. 2023 Jul;37(7):687-697. doi: 10.1177/02698811231179800. Epub 2023 Jun 30. PMID 37392016
- [Background] Anderson SM, Raghinaru D, Pinsker JE, Boscari F, Renard E, Buckingham BA, Nimri R, Doyle FJ 3rd, Brown SA, Keith-Hynes P, Breton MD, Chernavvsky D, Bevier WC, Bradley PK, Bruttomesso D, Del Favero S, Calore R, Cobelli C, Avogaro A, Farret A, Place J, Ly TT, Shanmugham S, Phillip M, Dassau E, Dasanayake IS, Kollman C, Lum JW, Beck RW, Kovatchev B; Control to Range Study Group. Multinational Home Use of Closed-Loop Control Is Safe and Effective. Diabetes Care. 2016 Jul;39(7):1143-50. doi: 10.2337/dc15-2468. Epub 2016 Apr 13. PMID 27208316
- [Background] Barba T, Buehler S, Kettner H, Radu C, Cunha BG, Nutt DJ, Erritzoe D, Roseman L, Carhart-Harris R. Effects of psilocybin versus escitalopram on rumination and thought suppression in depression. BJPsych Open. 2022 Sep 6;8(5):e163. doi: 10.1192/bjo.2022.565. PMID 36065128
- [Background] Carhart-Harris RL, Roseman L, Bolstridge M, Demetriou L, Pannekoek JN, Wall MB, Tanner M, Kaelen M, McGonigle J, Murphy K, Leech R, Curran HV, Nutt DJ. Psilocybin for treatment-resistant depression: fMRI-measured brain mechanisms. Sci Rep. 2017 Oct 13;7(1):13187. doi: 10.1038/s41598-017-13282-7. PMID 29030624
- [Background] Siegel JS, Subramanian S, Perry D, Kay BP, Gordon EM, Laumann TO, Reneau TR, Metcalf NV, Chacko RV, Gratton C, Horan C, Krimmel SR, Shimony JS, Schweiger JA, Wong DF, Bender DA, Scheidter KM, Whiting FI, Padawer-Curry JA, Shinohara RT, Chen Y, Moser J, Yacoub E, Nelson SM, Vizioli L, Fair DA, Lenze EJ, Carhart-Harris R, Raison CL, Raichle ME, Snyder AZ, Nicol GE, Dosenbach NUF. Psilocybin desynchronizes the human brain. Nature. 2024 Aug;632(8023):131-138. doi: 10.1038/s41586-024-07624-5. Epub 2024 Jul 17. PMID 39020167
- [Background] Zhao X, Du Y, Yao Y, Dai W, Yin Y, Wang G, Li Y, Zhang L. Psilocybin promotes neuroplasticity and induces rapid and sustained antidepressant-like effects in mice. J Psychopharmacol. 2024 May;38(5):489-499. doi: 10.1177/02698811241249436. Epub 2024 Apr 28. PMID 38680011
- [Background] Weleff J, Nunes JC, Costa GPA, Sofuoglu M, MacLean RR, De Aquino JP. From taboo to treatment: The emergence of psychedelics in the management of pain and opioid use disorder. Br J Clin Pharmacol. 2024 Dec;90(12):3036-3053. doi: 10.1111/bcp.16045. Epub 2024 Apr 16. PMID 38627909
- [Background] Shao LX, Liao C, Gregg I, Davoudian PA, Savalia NK, Delagarza K, Kwan AC. Psilocybin induces rapid and persistent growth of dendritic spines in frontal cortex in vivo. Neuron. 2021 Aug 18;109(16):2535-2544.e4. doi: 10.1016/j.neuron.2021.06.008. Epub 2021 Jul 5. PMID 34228959